CLINICAL TRIAL: NCT04768673
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety After Oral Administration of CKD-393 and Co-administration of CKD-501, D759 and H053 Under Fed Condition in Healthy Adults
Brief Title: A Study to Investigate the PK and Safety of CKD-393
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A98_04BE2022P
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-02

CONDITIONS: Type II Diabetes
Keywords: CKD-393; Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Period 1: CKD-501, D759, H053 / Period 2: CKD-393 Formulation I / Period 3: CKD-393 Formulation II
  Interventions: Drug: CKD-393 formulation I; Drug: CKD-393 formulation II; Drug: D501, D759, H053
- Group 2 (Experimental): Period 1: CKD-393 Formulation I / Period 2: CKD-393 Formulation II / Period 3: CKD-501, D759, H053
  Interventions: Drug: CKD-393 formulation I; Drug: CKD-393 formulation II; Drug: D501, D759, H053
- Group 3 (Experimental): Period 1: CKD-393 Formulation II / Period 2: CKD-501, D759, H053 / Period 3: CKD-393 Formulation I
  Interventions: Drug: CKD-393 formulation I; Drug: CKD-393 formulation II; Drug: D501, D759, H053
- Group 4 (Experimental): Period 1: CKD-501, D759, H053 / Period 2: CKD-393 Formulation II / Period 3: CKD-393 Formulation I
  Interventions: Drug: CKD-393 formulation I; Drug: CKD-393 formulation II; Drug: D501, D759, H053
- Group 5 (Experimental): Period 1: CKD-393 Formulation I / Period 2: CKD-501, D759, H053 / Period 3: CKD-393 Formulation II
  Interventions: Drug: CKD-393 formulation I; Drug: CKD-393 formulation II; Drug: D501, D759, H053
- Group 6 (Experimental): Period 1: CKD-393 Formulation II / Period 2: CKD-393 Formulation I / Period 3: CKD-501, D759, H053
  Interventions: Drug: CKD-393 formulation I; Drug: CKD-393 formulation II; Drug: D501, D759, H053

INTERVENTIONS:
Drug: CKD-393 formulation I — single, oral administration of 2 tablets under fed condition
Drug: CKD-393 formulation II — single, oral administration of 2 tablets under fed condition
Drug: D501, D759, H053 — single, oral administration of 1 D501, 1 D759 and 2 H053 under fed condition

SUMMARY:
A clinical trial to investigate the pharmacokinetics and safety after oral administration of CKD-393

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, two-way crossover clinical trial to investigate the pharmacokinetics and safety after oral administration of CKD-393 and co-administration of CKD-501, D759 and H053 under fed condition in healthy adults

ELIGIBILITY:
[Inclusion Criteria]

1. Between 19 aged and 50 aged healthy adult
2. Body weight more than 55kg for male, more than 50kg for female
3. Body Mass Index over 18.5kg/m2 and under 27.0kg/m2
4. if female, the subject must satisfy more than one of the following:

   * subject who have reached menopause (no natural menstruation for at least 2 years.)
   * subject who is surgically infertile(hysterectomy or bilateral salpingo-oophorectomy, tubal ligation, or in infertile state under other method)

[Exclusion Criteria]

1. Subject who is currently with or have diagnosed with clinically significant hepatobiliary(severe hepatopathy, etc.), kidney(severe nephropathy, etc.), neurological, immunologic, respiratory, urinary, gastrointestinal endocrinological(diabetic ketoacidosis, diabetic coma, etc.), hematological, oncological, cardiovascular(heart failure, etc.) or metal illness
2. Subject with one of the following laboratory test results

   * AST, ALT > UNLx1.5
   * eGRF < 60 ml/min/1.73 m2 (MDRD formula)
   * immuno-serology test results in positive
   * Systolic blood pressure > 150mmHg or <90mmHg, Diastolic blood pressure >100mmHg or <50mmHg
3. Subject who has history of the following and the history may affect safety of the subject or result of this study

   * History of any prescription drug or herbal medicine within 14 days before first administration investigational products
   * History of any non-prescription drug including health food, vitamin within 7 days before first administration investigational products
   * History of drug-metabolizing induction/inhibition enzyme such as barbital

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 h (hours), 0.25 h (hours), 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 24h, 32h, 48h
  Maximum concentration of drug in plasma
AUClast | 0 h (hours), 0.25 h (hours), 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 24h, 32h, 48h
  Area under the plasma drug concentration-time curve to last concentration

SECONDARY OUTCOMES:
AUCinf | 0 h (hours), 0.25 h (hours), 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 24h, 32h, 48h
  Area under the plasma drug concentration-time curve from 0 to infinity
Tmax | 0 h (hours)h, 0.25 h (hours), 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 24h, 32h, 48h
  Time to maximum plasma concentration
t1/2 | 0 h (hours), 0.25 h (hours), 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 24h, 32h, 48h
  Terminal elimination half-life
Vd/F | 0 h (hours), 0.25 h (hours)h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 24h, 32h, 48h
  Apparent Volume of Distribution
CL/F | 0 h (hours), 0.25 h (hours), 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 24h, 32h, 48h
  Apparent Clearance

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, MD, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu,, South Korea

IPD SHARING:
Plan to Share IPD: No